CLINICAL TRIAL: NCT04371718
Title: A Phase II, Randomized, Double-Blind, Placebo Controlled, Trial of JKB-122 as an Adjunct Therapy to Prednisolone and Azathioprine in the Induction of Remission in Autoimmune Hepatitis (AIH)
Brief Title: Effect of JKB-122 on Prednisolone and Azathioprine Induced Remission in Autoimmune Hepatitis (AIH)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TaiwanJ Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JKB-122 AIH01
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Autoimmune Hepatitis
Keywords: Autoimmune Hepatitis; Orphan Disease; Aminotransferase; Steroid sparing; ALT
MeSH Terms: conditions — Hepatitis, Autoimmune; Rare Diseases | interventions — JKB-122

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- JKB-122 Low dose (Experimental): JKB-122 5 mg daily for 104 weeks
  Interventions: Drug: JKB-122
- JKB-122 Medium dose (Experimental): JKB-122, 15 mg daily for 104 weeks
  Interventions: Drug: JKB-122
- JKB-122 High dose (Experimental): JKB-122 35 mg daily for 104 weeks
  Interventions: Drug: JKB-122
- Placebo (Placebo Comparator): Matched placebo, daily for 104 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JKB-122 — JKB-122 is a TLR antagonist to immune modulate for autoimmune hepatitis
  Arms: JKB-122 High dose; JKB-122 Low dose; JKB-122 Medium dose
Other: Placebo — A capsule has same component but active drug
  Arms: Placebo

SUMMARY:
This is a Phase 2 study. All patients will receive prednisolone and AZA as standard of care (SOC) during the study. At the end of the study, all data collected will be analyzed the efficacy and safety of JKB-122 on SOC reduction and inflammation improvement in Autoimmune Hepatitis

DETAILED DESCRIPTION:
JKB-122 has been demonstrated effective reducing aminotransferase in refractory AIH patients with SOC.This is a new Phase 2 study to find an optimal dose for relevant phase 3 study in newly diagnostic AIH patients. All patients will receive prednisolone and AZA as standard of care (SOC) during the study. Subjects will be randomized to receive 5 mg JKB-122, 15 mg JKB-122, 35 mg JKB-122 or placebo in 1:1:1:1 ratio, adjunct to SOC. This protocol with the primary endpoint being biochemical remission and evaluation of 3 different treatment doses. The histology will be explored as secondary to test long term benefit and to show similar trend with the biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 65 years old.
2. If female of childbearing potential, must not be pregnant or breastfeeding and either postmenopausal (no menses for previous 12 months) or using an effective method of birth control.
3. Probable or definite diagnosis of autoimmune hepatitis according to the International Autoimmune Hepatitis Study Group criteria.
4. New diagnosis of AIH that requires treatment according to the current EASL guidelines.
5. Has elevated liver test results (ALT) at least 5x ULN at screening.
6. Is capable of understanding and signing the informed consent document.

Exclusion Criteria:

1. Overlap syndrome with Primary Sclerosing Cholangitis (PSC) or Primary Biliary Cholangitis (PBC)
2. Has cirrhosis on liver biopsy, or Child-Pugh score greater than 6 at screening.
3. Has human immunodeficiency virus (HIV) or is hepatitis B virus or HCV positive.
4. Has history of alcohol intake > 25 g/day within the past six months.
5. Severe anemia, leukopenia , or thrombocytopenia.
6. Known intolerances to prednisolone or azathioprine.
7. Current treatment with prednisone/prednisolone and/or immunosuppressive medication for an indication other than autoimmune hepatitis
8. Has a known or suspected central nervous system disorder that may predispose to seizures or lower the seizure threshold
9. Has unstable and uncontrollable hypertension (>180/110 mmHg)
10. Has current malignancy or a history of malignancy (within the past 5 years), except basal or non-metastatic squamous cell carcinoma of the skin that has been treated successfully.
11. Has any form of current substance abuse, psychiatric disorder or a condition that, in the opinion of the Investigator, may invalidate communication with the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Reduction of inflammation in Autoimmune Hepatitis | 6, 12, and 24 months
  The % of patients in each treatment group who achieve biochemical remission

SECONDARY OUTCOMES:
Steroid sparing effect | week 104
  Steroid accumulation dose in overall or in those who achieve resolution of histology without worsening of the fibrosis
Changes in liver histology as measured by Hepatic Activity Index (HAI) | Week 104
  The reduction of inflammation in histology refers to improve Autoimmune Hepatitis disease status